CLINICAL TRIAL: NCT01332058
Title: Promoting Walking in African Americans With Peripheral Arterial Disease
Brief Title: Motivational Interviewing (MI) for African Americans With Peripheral Arterial Disease (PAD) Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tracie Collins, MD, MPH (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Tracie Collins, MD, MPH, Preventive Medicine and Public Health Chair, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R01HL09890901 - Pilot; R01HL098909 (NIH); 7R01HL098909-03 (NIH)
Record Dates: First submitted 2011-02-16; First posted 2011-04-08 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Walking; Motivational Interviewing
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — 8 possible weeks of motivational interviewing sessions

SUMMARY:
The investigators are conducting a pilot study for a clinical research trial to establish the feasibility and acceptability of the intervention and the most effective recruitment strategies prior to the full study.

DETAILED DESCRIPTION:
The eight week pilot will be conducted to establish the feasibility of implementing motivational interviewing as a means to counsel African Americans with peripheral arterial disease (PAD) to increase their walking. Additionally, we will determine the acceptance of culturally sensitive print material on managing PAD. Finally, we will utilize the pilot to develop best practice methods for successfully carrying out the full study.

ELIGIBILITY:
Inclusion Criteria:

* African American (determined by self-report)
* Lived most of their life in the United States
* Resting ABI <0.95
* English Speaking
* Has a telephone

Exclusion Criteria:

* Currently walking for exercise at least 5 days per week (i.e., a PACE score ranging from 5-8)
* Prior major amputation (foot or lower leg) or critical leg ischemia (tissue loss, gangrene, or ulcers)
* Rest pain with ABI <0.4 and non-palpable femoral pulses without prior evaluation by a vascular surgeon, given the need for evaluation for the role of more invasive therapy prior to recommending walking therapy
* Leg revascularization within 3 months of enrollment or plans for revascularization during the study period
* Use of supplemental oxygen
* Myocardial infarction within the preceding 3 months
* Resting blood pressure > 200/110 mmHg
* Exercise-induced coronary ischemic symptoms, or exercise-induced ST depression > 2.0 mm
* Inability to walk for 2 minutes; the rationale being that people who cannot walk for 2 minutes would not be able to complete the necessary submaximal treadmill test, which is used to screen for coronary ischemic symptoms. We will also exclude anyone who can walk for 20 minutes or more during the submaximal treadmill test. Anyone who can complete the submaximal test would not have significant walking impairment and would not get that much out of the study.
* Short Physical Performance Battery score of 10 or higher as such persons do not have a clinically significant impairment in mobility; therefore, we will exclude anyone who scores a 10 or higher (out of a maximum of 12 points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to eight weeks in 6 minute walk test | 8 weeks
  The participant will walk as far as possible for 6 minutes in a marked corridor. They will be permitted to slow down, stop, and to rest as necessary, but the time will continue to run. They will be given standardized encouragement at each minute and their ending point will be marked with tape. The laps will be counted and the total distance in feet will be recorded. The onset of claudication, number of times the participant needed to stop, and rate of perceived exertion will be recorded throughout the test.

SECONDARY OUTCOMES:
Baseline six minute walk test | baseline
  The participant will walk as far as possible for 6 minutes in a marked corridor. They will be permitted to slow down, stop, and to rest as necessary, but the time will continue to run. They will be given standardized encouragement at each minute and their ending point will be marked with tape. The laps will be counted and the total distance in feet will be recorded. The onset of claudication, number of times the participant needed to stop, and rate of perceived exertion will be recorded throughout the test.
Baseline 7 day physical activity | baseline
  Each participant will wear an accelerometer for one week at baseline to collect their current level physical activity. The accelerometers will collect movement in x, y, and z axis as well as total steps. They will be asked to put the accelerometer on first thing in the morning and take it right before bed.
Change from baseline to eight weeks 7 day physical activity | 8 weeks
  Each participant will wear an accelerometer for one week at baseline to collect their current level physical activity. The accelerometers will collect movement in x, y, and z axis as well as total steps. They will be asked to put the accelerometer on first thing in the morning and take it right before bed.

CONTACTS AND LOCATIONS:
Overall Officials: Tracie C Collins, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Wichita, Kansas, United States